CLINICAL TRIAL: NCT03415347
Title: De-roofing and Curettage Versus Wide Local Excision for the Treatment of Acute Pilonidal Abscess: A Randomised Controlled Trial
Brief Title: De-roofing and Curettage vs WLE for Pilonidal Abscess
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 241937
Record Dates: First submitted 2018-01-19; First posted 2018-01-30 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-01

CONDITIONS: Pilonidal Abscess; Pilonidal Sinus With Abscess; Pilonidal Sinus Infected; Pilonidal Disease
Keywords: Pilonidal abscess; Pilonidal disease; Pilonidal sinus
MeSH Terms: conditions — Pilonidal Sinus | interventions — Curettage

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of two groups, intervention 1 (abscess de-roofing and curettage) or intervention 2 (abscess wide local excision), then followed up for 1 year to detect recurrence rate of pilonidal abscess
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abscess de-roofing and curettage (Active Comparator): Abscess de-roofing and curettage. The patient will be placed in the lateral position with the buttocks spread apart using tape. The cleft of the buttocks will be shaved prior to cleaning and preparation of the skin. A spindle-shaped (elliptical) excision will be performed to the lateral aspect of the abscess formation with a scalpel staying away from the midline. Once the pus has been drained through this lateral incision the wound cavity will then be curetted and washed out with hydrogen peroxide. The wound size will be measured by the operating surgeon who will record the maximal length and width of the wound. Once haemostasis (cessation of any bleeding) is achieved the wound will be packed with Kaltostat ribbon and the wound dressed with blue gauze and mefix tape. The wound is therefore left open.
  Interventions: Procedure: Abscess de-roofing and curettage
- Abscess wide local excision (Active Comparator): Wide local excision. Patients will be placed in the prone position with the buttocks spread apart using tape. The cleft of the buttocks will be shaved prior to cleaning and preparation of the skin. Diluted methylene blue will be injected in all visible pits and a wide spindle-shaped (elliptical) midline excision of the skin and the underlying subcutaneous tissue down to the coccygeal (pre-sacral) fascia including all sinuses will be performed with electrocautery. The specimen will be sent for histology as per routine surgical practice. The wound will be washed with hydrogen peroxide. The wound size will be measured by the operating surgeon who will record the maximal length and width of the wound. Once haemostasis (cessation of any bleeding) is achieved the wound will be packed with Kaltostat ribbon and the wound dressed with blue gauze and mefix tape. The wound is therefore left open.
  Interventions: Procedure: Abscess wide local excision

INTERVENTIONS:
Procedure: Abscess de-roofing and curettage — Abscess de-roofing and curettage
  Arms: Abscess de-roofing and curettage
Procedure: Abscess wide local excision — Abscess wide local excision
  Arms: Abscess wide local excision

SUMMARY:
Pilonidal disease refers to a common disease affecting mostly young males. It may present as asymptomatic pits, acute and painful abscess formation, or chronic discharging sinuses. There are many treatment options for the latter two manifestations but broadly speaking the surgical treatment of acute pilonidal abscess can fall into three categories: (1) incision and drainage, (2) de-roofing and curettage and (3) wide local excision.

The evidence available for the surgical management of acute pilonidal abscess is limited. Previous studies have consistently demonstrated that incision and drainage results in high recurrence rates and should not be considered as the first-line treatment option for the management of acute pilonidal abscess. However, it is not clear whether abscess de-roofing with curettage or wide local excision should be considered as the surgical procedure of choice in acute pilonidal abscess. There has not been a prospective randomised study comparing abscess de-roofing with curettage and wide local excision for acute pilonidal abscess. The ideal surgical procedure would be one that results in the lowest rate of abscess recurrence, treats the underlying pilonidal sinus thereby reducing the need for re-operation but has acceptable post-operative pain, complications and time to complete wound healing.

DETAILED DESCRIPTION:
BACKGROUND

Pilonidal disease refers to a common disease affecting mostly young males. It may present as asymptomatic pits, acute and painful abscess formation, or chronic discharging sinuses. There are many treatment options for the latter two manifestations but broadly speaking the surgical treatment of acute pilonidal abscess can fall into three categories: (1) incision and drainage, (2) de-roofing and curettage and (3) wide local excision.

Some authors believe that the incision and drainage method is an effective procedure. However, this method would treat only the acute infection and produce the necessity of re-operation for definite therapy. The alternative method is wide local excision in which the patients receive definite therapy in a single staged operation reducing the number of operations per patient, patient visits to hospital and overall cost to the health service. However, concerns over the length of time to gain acceptable wound healing following wide local excision has decreased its popularity with some surgeons. There is limited evidence available for the surgical management of acute pilonidal abscess which has lead to disagreement as to what is the best option. One randomised study of 76 patients compared incision and drainage of acute pilonidal abscess followed by an elective excision of the pilonidal sinus and primary closure at 3 weeks versus wide local excision with the wound left open for secondary healing. At 12 months the incision and drainage followed by elective excision group had 14% recurrence of pilonidal abscess whereas the wide local excision group had 0% recurrence. Another randomised study of 131 patients compared incision and drainage versus abscess excision (de-roofing) with curettage for acute pilonidal abscess and found recurrence rates of 42% in the incision and drainage group verses 11% in the curettage group. A prospective randomised study similarly compared incision and drainage versus abscess excision (de-roofing) with curettage for acute pilonidal abscess and reported a significantly higher rate of developing a chronic pilonidal sinus in the incision and drainage group (76% vs 24%, p<0.001). A retrospective study with median follow up of 5.3 years has recently been published comparing abscess de-roofing with curettage and wide local excision for acute pilonidal abscess. The authors reported an approximate three-fold increase in recurrence rate in the curettage group compared with the wide local excision group.

RATIONALE FOR CURRENT STUDY

The evidence available for the surgical management of acute pilonidal abscess is limited. Previous studies have consistently demonstrated that incision and drainage results in high recurrence rates and should not be considered as the first-line treatment option for the management of acute pilonidal abscess. However, it is not clear whether abscess de-roofing with curettage or wide local excision should be considered as the surgical procedure of choice in acute pilonidal abscess. There has not been a prospective randomised study comparing abscess de-roofing with curettage and wide local excision for acute pilonidal abscess. The ideal surgical procedure would be one that results in the lowest rate of abscess recurrence, treats the underlying pilonidal sinus thereby reducing the need for re-operation but has acceptable post-operative pain, complications and time to complete wound healing.

Research question:

Does wide local excision when compared to abscess excision (de-roofing) with curettage result in reduced recurrence rates and therefore provide a single-stage procedure for the management of acute pilonidal abscess and the underlying causative sinus? Is wide local excision when compared to abscess de-roofing with curettage a safe procedure in terms of complications (bleeding, wound infection), post-operative pain and time to complete wound healing?

Hypothesis:

Wide local excision for the management of acute pilonidal abscess results in lower recurrence rates when compared with abscess de-roofing with curettage. Post-operative pain, complications and time to complete wound healing will not be significantly different between the two treatment groups.

STUDY OBJECTIVES

Primary objectives:

To compare therapeutic values of abscess de-roofing with curettage versus wide local excision in the surgical treatment of patients with acute pilonidal abscess. Therapeutic values include: recurrence rate, post-operative pain, time to complete wound healing, time to returning to work or normal daily activities and complications of surgery (bleeding and wound infection).

Secondary objectives:

To assess the practicality of abscess de-roofing with curettage and wide local excision in the surgical treatment of patients with acute pilonidal abscess in terms of operative time and total time in theatre.

STUDY DESIGN

Type of study: Single centre randomised controlled clinical trial

Study design:

Patients with acute pilonidal abscess will be randomised into 2 treatment groups. Randomisation of patients will be performed by the surgical registrar on call for either admissions or the emergency theatre. The method of randomisation will be by identical sealed envelopes. The principle investigator (Lalin Navaratne) will create trial packs within identical sealed envelopes. These packs will contain:

1. Patient information sheet (PIS)
2. 3 copies of the patient consent form (for the study)
3. A consent form for the operation (Consent Form 1)
4. Information sheet to the operating surgeon outlining which treatment arm the patient has been allocated to
5. The data collection sheet(s) for demographic data, medical history, smoking history, previous pilonidal disease history, operative data, and follow up data
6. Letter to GP

The sealed envelopes will be created in blocks of 20 (10 for each treatment arm) to keep the groups of similar size during the study. Once the 20 envelopes have been created and sealed (with a signed white label) they will be shuffled by another investigator who has not been involved in creating the packs and placed in a secure location (locked filing cabinet within the surgical assessment unit). When a patient has been referred to the emergency surgery unit they will be seen on the surgical assessment unit and will be invited to join the study if inclusion and exclusion criteria have been met. The patient will be given the Patient Information Sheet (PIS) and have adequate time to read it. Once the patient has read the PIS and had an opportunity to ask any questions they will be enrolled into the study if applicable. The surgeon will take the trial pack 'on the top of the pile' within the secured filing cabinet which will randomly allocate the patient to one of two treatment arms. The two treatment arms are: (1) de-roofing and curettage and (2) wide local excision. The surgeon will complete any data collection requirements at this stage and all documentation will remain in the envelope and be tracked with the patients notes.

The two arms of this trial will be performed in the operating theatre with the patient under general anaesthesia. The surgical technique for each treatment arm is detailed below:

1. Abscess de-roofing and curettage. The patient will be placed in the lateral position with the buttocks spread apart using tape. The cleft of the buttocks will be shaved prior to cleaning and preparation of the skin. A spindle-shaped (elliptical) excision will be performed to the lateral aspect of the abscess formation with a scalpel staying away from the midline. Once the pus has been drained through this lateral incision the wound cavity will then be curetted and washed out with hydrogen peroxide. The wound size will be measured by the operating surgeon who will record the maximal length and width of the wound. Once haemostasis (cessation of any bleeding) is achieved the wound will be packed with Kaltostat ribbon and the wound dressed with blue gauze and mefix tape. The wound is therefore left open.
2. Wide local excision. Patients will be placed in the prone position with the buttocks spread apart using tape. The cleft of the buttocks will be shaved prior to cleaning and preparation of the skin. Diluted methylene blue will be injected in all visible pits and a wide spindle-shaped (elliptical) midline excision of the skin and the underlying subcutaneous tissue down to the coccygeal (pre-sacral) fascia including all sinuses will be performed with electrocautery. The specimen will be sent for histology as per routine surgical practice. The wound will be washed with hydrogen peroxide. The wound size will be measured by the operating surgeon who will record the maximal length and width of the wound. Once haemostasis (cessation of any bleeding) is achieved the wound will be packed with Kaltostat ribbon and the wound dressed with blue gauze and mefix tape. The wound is therefore left open.

Patients will not be routinely prescribed any antibiotics following the operation. All patients will have wound packing for the first 24 hours after the operation. For patients within the drainage and curettage group no further packing is usually required. Patients discharged the same day of surgery will have their packing removed and wound reviewed in the community. Patients who stay in-hospital overnight following their surgery will have their packing removed and wound reviewed in-hospital prior to discharge. For patients within the wide local excision group, packing may be required following the first post-operative day and packing is continued until no longer indicated. Dressing changes for these patients will occur in the community.

All patients will be advised to cleanse the wounds in the shower at least once a day and will be followed up in a dedicated wound clinic weekly until their wounds have healed. After healing, they will be followed up in a telephone clinic at 6 and then 12 months. When attending the wound clinic, data will be collected on abscess recurrence, time to wound healing, number of days until the patient can return to work (or when they resumed normal daily activities), pain scores, wound size and any signs of wound infection. Further follow up in the main outpatient department will monitor for abscess recurrence. With patient consent, non-identifying photographs may be taken of the wound during the operation and the subsequent healing process during the follow up period.

Any patient enrolled within the study may re-present with an acute abscess recurrence within the follow up period of one year. If the patient belongs to the de-roof and curettage group, they would be offered a wide local excision as the surgical management of choice. If the patient belongs to the wide local excision group, then they would be offered further drainage and curettage or wide local excision based on what the attending surgeon feels is the best surgical option for that particular patient. Analysis would be by intention to treat. Any patient re-operated on during the study period would not need to be followed up in the weekly wound clinic for the purposes of data collection (time to healing, time to returning to work, pain scores, wound size etc). These patients would be followed up in the outpatient clinic as per departmental standard operating procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute pilonidal abscess

Exclusion Criteria:

* Patients under the age of 16 years will be excluded.
* Immunocompromised (diabetes mellitus, taking oral steroids or immunosuppressive medication) patients will be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pilonidal abscess | 1 year
  During the follow up period the primary outcome measure will be if the patient develops a (recurrent) pilonidal abscess. This is a clinical diagnosis made by the clinician (General Practitioner or Hospital Doctor) attending to the patient. The definition for recurrent pilonidal abscess is any pilonidal abscess that occurs requiring either antibiotic (oral or intravenous) or surgical treatment. A small amount of discharge that settles on its own without the need for such treatment will not be counted as a recurrence.

SECONDARY OUTCOMES:
Time to complete wound healing | 4-10 weeks
  Defined as not requiring any further wound dressings
Return to work | 2-8 weeks
  Number of days until returning to work (if unemployed then number of days until resuming normal daily activities)
Procedural time | 1 hour
  Operative time and total time in theatre
Wound size at operation | 1 hour
  Maximal length and width in cm)
Wound size over time | 4-10 weeks
  Maximal length and width in cm weekly until wound healed
Post-operative pain scores | 4-10 weeks
  Using a visual analogue scale weekly until wound healed
Patient wound impact questionnaire | 4-10 weeks
  Cardiff Wound Impact Questionnaire to be performed on the first and last weekly wound review clinic
Wound infection rate | 4-10 weeks
  Infection during the wound healing phase that requires any form of antibiotic (topical, oral or intravenous)

CONTACTS AND LOCATIONS:
Overall Officials: Lalin Navaratne, MBBS MRCS, Principal Investigator — LONDON NORTH WEST UNIVERSITY HEALTHCARE NHS TRUST

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loganathan A, Arsalani Zadeh R, Hartley J. Pilonidal disease: time to reevaluate a common pain in the rear! Dis Colon Rectum. 2012 Apr;55(4):491-3. doi: 10.1097/DCR.0b013e31823fe06c. No abstract available. PMID 22426275
- [Background] Hosseini SV, Bananzadeh AM, Rivaz M, Sabet B, Mosallae M, Pourahmad S, Yarmohammadi H. The comparison between drainage, delayed excision and primary closure with excision and secondary healing in management of pilonidal abscess. Int J Surg. 2006;4(4):228-31. doi: 10.1016/j.ijsu.2005.12.005. Epub 2006 May 22. PMID 17462356
- [Background] Vahedian J, Nabavizadeh F, Nakhaee N, Vahedian M, Sadeghpour A. Comparison between drainage and curettage in the treatment of acute pilonidal abscess. Saudi Med J. 2005 Apr;26(4):553-5. PMID 15900358
- [Background] Eryilmaz R, Sahin M, Alimoglu O, Kaya B. [The comparison of incision and drainage with skin excision and curettage in the treatment of acute pilonidal abscess]. Ulus Travma Acil Cerrahi Derg. 2003 Apr;9(2):120-3. Turkish. PMID 12836108
- [Background] Fahrni GT, Vuille-Dit-Bille RN, Leu S, Meuli M, Staerkle RF, Fink L, Dincler S, Muff BS. Five-year Follow-up and Recurrence Rates Following Surgery for Acute and Chronic Pilonidal Disease: A Survey of 421 Cases. Wounds. 2016 Jan;28(1):20-6. PMID 26824973